CLINICAL TRIAL: NCT04745767
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Relative Bioavailability of Different TAK-994 Formulations and the Effect of Food on These Formulations in Healthy Adult Subjects
Brief Title: A Study of Different Forms of TAK-994 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TAK-994-1006
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Healthy Participants
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: A1(T1), B(T2), C(T2 Fed) (Experimental): Participants will be randomly placed into 6 sequences within Group 1. All participants in Group 1 will receive TAK-994 as Treatment A1 (T1 Formulation) and Treatment B (T2 Formulation) under fasted conditions and Treatment C (T2 Formulation) under fed conditions at different times within three periods.
  Interventions: Drug: TAK-994
- Group 2: A2(T1), D(T3), E(T3 Fed) (Experimental): Participants will be randomly placed into 6 sequences within Group 2. All participants in Group 2 will receive TAK-994 as Treatment A2 (T1 Formulation) and Treatment D (T3 Formulation) under fasted conditions and Treatment E (T3 Formulation) under fed conditions at different times within three periods.
  Interventions: Drug: TAK-994
- Group 3: A3(T1), F(T4), G(T4 Fed), H(T5) (Experimental): Participants will be randomly placed into 6 sequences within Group 3. Participants in Group 3 will receive TAK-994 as Treatment A3 (T1 Formulation), Treatment F (T4 Formulation), and Treatment F (T5 Formulation) under fasted conditions and Treatment G (T4 Formulation) under fed conditions at different times within 4 periods.
  Interventions: Drug: TAK-994

INTERVENTIONS:
Drug: TAK-994 — T2 formulation.
  Arms: Group 1: A1(T1), B(T2), C(T2 Fed)
Drug: TAK-994 — T1 formulation.
Drug: TAK-994 — T3 formulation.
  Arms: Group 2: A2(T1), D(T3), E(T3 Fed)
Drug: TAK-994 — T4 formulation.
  Arms: Group 3: A3(T1), F(T4), G(T4 Fed), H(T5)
Drug: TAK-994 — T5 formulation.
  Arms: Group 3: A3(T1), F(T4), G(T4 Fed), H(T5)

SUMMARY:
It is hoped that TAK-994 will eventually help people with a sleep condition called narcolepsy. Narcolepsy is a condition that causes extreme sleepiness during the day, including falling asleep suddenly. Before then, the sponsor needs to understand how the body processes TAK-994.

The main aims of the study are to learn how the body processes 4 different new forms of TAK-994, when taken with food and without food, compared to a standard form of TAK-994.

At the first visit, the study doctor will check who can take part. Then the participants will be picked for 1 of 3 groups by chance. These groups of participants will take different new forms of TAK-994 and the standard form. They will take these with and without food. This will happen again 3 or 4 times but will take TAK-994 in a different order each time. After each treatment with TAK-994, the study doctors will check the amount of TAK-994 in the blood of the participants, over time. The study doctors will also check if the participants have any side effects from TAK-994.

Participants will wait 5 or more days between each dose to allow time for TAK-994 to completely leave their bodies. Participants will stay in the clinic during their treatment with TAK-994. They will stay in the clinic for 15 days or longer. Participants who have 4 treatments with TAK-994 will stay in the clinic for 20 days or longer.

Then, the clinic will telephone the participants 12 days after their final treatment of TAK-994 to check if they have any health problems.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-994. TAK-994 is being tested in healthy participants. This study will look at the relative BA of different TAK-994 test formulations relative to the currently used formulation (T1) and the effect of food on the test formulations in healthy participants.

The study will enroll approximately 54 participants. The study consists of three parallel groups (Group 1, Group 2, and Group 3). In each group, one test TAK-994 formulation (T2 formulations in Group 1; T3 formulations in Group 2; and T4 and T5 formulations in Group 3) will be evaluated under fed and fasting condition compared to reference T1 formulation under fasting conditions in a cross-over design. Participants will be randomly assigned into 6 sequences within each group.

This multi-center trial will be conducted in United States. The overall time to participate in this study is approximately 57 days. Participants will be followed up for up to 14 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilogram per square meter (kg/m^2) at the screening.
2. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator or designee.

Exclusion Criteria:

1. Mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. Current or past history of epilepsy, seizure, or convulsion, tremor, or related symptoms.
3. Positive urine drug or alcohol results at screening or check-in.
4. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
5. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine), of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
6. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
7. Is lactose intolerant or unable/unwilling to eat the high-fat/high-calorie breakfast.
8. Donation of blood or significant blood loss within 56 days prior to the first dosing.
9. Plasma donation within 7 days prior to the first dosing.
10. Participation in another clinical study within 30 days or 5 half-lives (whichever is longer) prior to the first dosing. The 30-day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Cmax : Maximum Observed Plasma Concentration for TAK-994 | Day 1: Pre-dose and at multiple time points (up to 72 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-994 | Day 1: Pre-dose and at multiple time points (up to 72 hours) post-dose
AUC∞: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for TAK-994 | Day 1: Pre-dose and at multiple time points (up to 72 hours) post-dose

SECONDARY OUTCOMES:
Number of Participants With at Least one Treatment-emergent Adverse Event (TEAE) | Day 1 up to 14 days after last dose of study drug (up to Day 33)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Celerion Tempe, AZ site, Tempe, Arizona
  - Celerion Lincoln, NE site, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/6026b26c5f53e3001ed0d7d3